CLINICAL TRIAL: NCT03665454
Title: A Phase Ib Safety, Tolerability, and Efficacy Study of Two Days of Oral Split Dose (25/20 mg) Administration of PF 06412562 in Subjects With Advanced Stage Parkinson's Disease
Brief Title: PF 06412562 in Subjects With Advanced Stage Parkinson's Disease
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Milton S. Hershey Medical Center (Other)
Collaborators: Pfizer (Industry)
Responsible Party: Principal Investigator, Xuemei Huang, MD, PhD, Professor, Department of Neurology, Milton S. Hershey Medical Center
Allocation: Randomized | Model: Crossover | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 9437
Record Dates: First submitted 2018-08-01; First posted 2018-09-11 (Actual); Last update posted 2019-07-31 (Actual); Status verified 2019-07

CONDITIONS: Parkinson Disease
Keywords: Parkinson's Disease; Parkinson Disease; End-Stage; Progressed; Advanced Parkinson's Disease; End-Stage Parkinson's Disease; Clinical intervention; Double-blind, randomized
MeSH Terms: conditions — Parkinson Disease | interventions — carbidopa, levodopa drug combination

STUDY DESIGN:
Intervention Model Description: Subjects will participate in study for 2 consecutive weeks. Days 2-3 of Week 1, they will be blindly and randomly assigned to one of two treatment arms (study drug PF-06412562 or standard of care carbidopa/levodopa). Whichever treatment arm they did not receive during Week 1, they will receive during Days 2-3 of Week 2.
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Masking Description: Investigational Drug Services, which is the investigational drug pharmacy at Hershey Medical Center, will be preparing and dispensing the drug. They will be the only party that is unblinded. Pfizer will provide placebo pills that are identical in appearance to the PF-06412562 study drug. The standard of care treatment, carbidopa/levodopa, is different in appearance to PF-06412562 and its corresponding matching placebo. In order to blind for this, Investigational Drug Services will encapsulate the carbidopa/levodopa pills. Thus, subjects may receive either an encapsulated carbidopa/levodopa pill or an empty non-active capsule, depending on the treatment arm and dosing they are scheduled to receive.
Oversight: FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- PF-06412562 (Experimental): Subjects will receive 25 mg of PF-06412562 twice daily on study Days 2 and 3, along with placebo carbidopa/levodopa dosed at these times. Additional carbidopa/levodopa placebo capsules also will be administered according to the subject's home regimen.
  Interventions: Drug: PF-06412562
- Standard of Care carbidopa/levodopa (Active Comparator): Subjects will take placebo tablets for the PF-06412562 twice daily on study Days 2 and 3, along with active carbidopa/levodopa (25/100 mg) administered at these times. Additional active carbidopa/levodopa capsules also will be administered according to the subject's home regimen.
  Interventions: Drug: Standard of Care Placebo

INTERVENTIONS:
Drug: PF-06412562 — PF-06412562 is a dopamine agonist developed by Pfizer Inc. into a tablet form for oral usage. It will be provided as 5 mg tablets. Thus, to administer the 25 mg dose, 5 x 5 mg tablets will be given; and to administer the 20 mg dose, 4 x 5 mg tablets will be administered.
  Arms: PF-06412562
Drug: Standard of Care Placebo — 25/100 mg tablet(s) of carbidopa/levodopa will be encapsulated and administered according to the subject's home regimen.
  Other Names: Sinemet
  Arms: Standard of Care carbidopa/levodopa

SUMMARY:
The purpose of this study is to test the safety and tolerability of the investigational drug PF-06412562 compared to the current medical standard of care medication for Parkinson's disease, carbidopa/levodopa. This research also is being done to find out if the investigational drug PF-06412562 can help improve the motor (movement) function, alertness, and cognitive (thinking) skills of people who are considered to be in the advanced-stage of Parkinson's disease. In this study, PF06412562 is 'investigational,' which means that it is experimental and has not been approved by the US Food and Drug Administration (FDA), but can be used in clinical research studies such as this one.

DETAILED DESCRIPTION:
The investigators are conducting a randomized, double-blind, carbidopa/levodopa-controlled crossover safety, tolerability, and efficacy study of the investigational compound, PF-06412562, in advanced Parkinson's patients. The primary purpose of this study is to test the safety and tolerability of the investigational drug PF-06412562 compared to the current medical standard of care medication for Parkinson's disease, carbidopa/levodopa, in these patients. This secondary purpose of this research is to find out if the investigational drug PF-06412562 can help improve the motor (movement) function, alertness, and cognitive (thinking) skills of people who are considered to be in the advanced-stage of Parkinson's disease. This study will inform the field as to whether PF-06412562 is safe and well-tolerated in advanced Parkinson's patients, and also may provide preliminary data on its efficacy in several domains.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of classic PD with history of clinically meaningful response to levodopa
* Disease duration >15 years since diagnosis
* Hoehn & Yahr stage >IV "on" or "off" levodopa
* Consent signed by subject, if possible
* If subject is cognitively impaired, consent signed by power of attorney or legally authorized subject representative
* Assent from the study subject, if possible
* Stable dose of all medications for 60 days prior to Day 1 of first week of study

Exclusion Criteria:

* Atypical parkinsonian syndrome (e.g., never responded to levodopa, and/or atypical signs)
* Acute or unstable medical condition such as heart disease, kidney and liver failure
* History of HIV, hepatitis B and C
* Use of moderate to strong CYP 3A4 modulators (see both inhibitors and inducers in Appendix BB)

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 8 (Actual)
Dates: Start 2018-09-24 (Actual); Primary Completion 2019-03-21 (Actual); Study Completion 2019-04-21 (Actual)

PRIMARY OUTCOMES:
Safety and tolerability of PF-06412562 assessed by blood sample results | Day 1
  NA (mmol/L), K(mmol/L), HCO3(mmol/L)
Safety and tolerability of PF-06412562 assessed by blood sample results | Day 1
  Ca (mg/dL), Mg (mg/dL), BUN( mg/dL), Creatinine (mg/dL), Bilirubin (mg/dL)
Safety and tolerability of PF-06412562 assessed by blood sample results | Day 1
  AST (U/L), ALT (U/L)
Safety and tolerability of PF-06412562 assessed by blood sample results | Day 1
  white blood cell count (K/uL), platelets (K/uL)
Safety and tolerability of PF-06412562 assessed by blood sample results | Day 1
  Hematocrit (%)
Safety and tolerability of PF-06412562 assessed by blood sample results | Day 1
  hemoglobin (g/dL)
Safety and tolerability of PF-06412562 assessed by blood sample results | Day 4
  NA (mmol/L), K(mmol/L), HCO3(mmol/L)
Safety and tolerability of PF-06412562 assessed by blood sample results | Day 4
  Ca (mg/dL), Mg (mg/dL), BUN (mg/dL), creatinine (mg/dL), bilirubin (mg/dL)
Safety and tolerability of PF-06412562 assessed by blood sample results | Day 4
  AST (U/L), ALT (U/L)
Safety and tolerability of PF-06412562 assessed by blood sample results | Day 4
  white blood cell count (K/uL), platelets (K/uL)
Safety and tolerability of PF-06412562 assessed by blood sample results | Day 4
  hematocrit (%)
Safety and tolerability of PF-06412562 assessed by blood sample results | Day 4
  hemoglobin (g/dL)
Safety and tolerability of PF-06412562 assessed by blood sample results | Day 4
  Red blood cell count (M/uL)
Safety and tolerability of PF-06412562 assessed by vital signs | Time Frame: Vital signs: X2 on Day 1
  height (inches)
Safety and tolerability of PF-06412562 assessed by vital signs | X2 on Day 1
  weight (lbs)
Safety and tolerability of PF-06412562 assessed by vital signs | X2 on Day 1
  blood pressure (mmHg)
Safety and tolerability of PF-06412562 assessed by vital signs | X2 on Day 1
  heart rate (bpm)
Safety and tolerability of PF-06412562 assessed by vital signs | X2 on Day 1
  respiratory rate (breathes/min)
Safety and tolerability of PF-06412562 assessed by vital signs | X2 on Day 1
  temperature (F)
Safety and tolerability of PF-06412562 assessed by vital signs | X3 on Days 2
  height (inches)
Safety and tolerability of PF-06412562 assessed by vital signs | X3 on Days 2
  blood pressure (mmHg)
Safety and tolerability of PF-06412562 assessed by vital signs | X3 on Days 2
  heart rate (bpm)
Safety and tolerability of PF-06412562 assessed by vital signs | X3 on Days 2
  respiratory rate (breathes/min)
Safety and tolerability of PF-06412562 assessed by vital signs | X3 on Days 2
  temperature (F)
Safety and tolerability of PF-06412562 assessed by vital signs | X3 on Days 3
  height (inches)
Safety and tolerability of PF-06412562 assessed by vital signs | X3 on Days 3
  weight (lbs)
Safety and tolerability of PF-06412562 assessed by vital signs | X3 on Days 3
  blood pressure (mmHg)
Safety and tolerability of PF-06412562 assessed by vital signs | X3 on Days 3
  heart rate (bpm)
Safety and tolerability of PF-06412562 assessed by vital signs | X3 on Days 3
  respiratory rate (breathes/min)
Safety and tolerability of PF-06412562 assessed by vital signs | X3 on Days 3
  temperature (F)
Safety and tolerability of PF-06412562 assessed by vital signs | X2 on Day 4
  height (inches)
Safety and tolerability of PF-06412562 assessed by vital signs | X2 on Day 4
  weight (lbs)
Safety and tolerability of PF-06412562 assessed by vital signs | X2 on Day 4
  blood pressure (mmHg)
Safety and tolerability of PF-06412562 assessed by vital signs | X2 on Day 4
  heart rate (bpm)
Safety and tolerability of PF-06412562 assessed by vital signs | X2 on Day 4
  respiratory rate (breathes/min)
Safety and tolerability of PF-06412562 assessed by vital signs | X2 on Day 4
  temperature (F)
Safety and tolerability of PF-06412562 assessed by cardiology testing/cardiac autonomic function | X1 on Day 1 over 15 min
  Blood pressure (mmHg), cold pressor test measuring blood pressure (mmHg)
Safety and tolerability of PF-06412562 assessed by cardiology testing/cardiac autonomic function | X1 on Day 1 over 15 min
  heart rate (beats/min), sinus arrhythmia (beats/min)
Safety and tolerability of PF-06412562 assessed by cardiology testing/cardiac autonomic function | X3 on Days 2 over 15 min each time
  Blood pressure (mmHg), cold pressor test measuring blood pressure (mmHg)
Safety and tolerability of PF-06412562 assessed by cardiology testing/cardiac autonomic function | X3 on Days 2 over 15 min each time
  heart rate (beats/min), sinus arrhythmia (beats/min)
Safety and tolerability of PF-06412562 assessed by cardiology testing/cardiac autonomic function | X3 on Days 3 over 15 min each time
  Blood pressure (mmHg), cold pressor test measuring blood pressure (mmHg)
Safety and tolerability of PF-06412562 assessed by cardiology testing/cardiac autonomic function | X3 on Days 3 over 15 min each time
  heart rate (beats/min), sinus arrhythmia (beats/min)
Safety and tolerability of PF-06412562 assessed by UPDRS-IV | X3 on Days 2
  UPDRS-IV (United Parkinson's Disease Rating Scale): each questions scored on scale of 0 to 4, where 0= not present, 4= severe; subscales are summed to yield a total score, min total score:0, max total score:81; higher score corresponds to increased disease severity
Safety and tolerability of PF-06412562 assessed by UPDRS-IV | X3 on Days 3
  UPDRS-IV (United Parkinson's Disease Rating Scale): each questions scored on scale of 0 to 4, where 0= not present, 4= severe; subscales are summed to yield a total score, min total score:0, max total score:81; higher score corresponds to increased disease severity
Safety and tolerability of PF-06412562 assessed by Columbia Suicide Rating | X1 on Day 1
  C-SSRS measures suicidal ideation and/or behavior. Rated from Category 1-10 with Category 1 being the least severe, and Category 10 representing the most severe, i.e. completing suicide.
Safety and tolerability of PF-06412562 assessed by Columbia Suicide Rating | X1 on Day 4
  C-SSRS measures suicidal ideation and/or behavior. Rated from Category 1-10 with Category 1 being the least severe, and Category 10 representing the most severe, i.e. completing suicide.

SECONDARY OUTCOMES:
Pilot data on potential efficacy of PF-06412562 compared to the standard of care treatment (i.e., carbidopa/levodopa) on overall signs and quality of life in subjects with advanced PD | Global Impression of Change: X3 on Days 2 and 3; Caregiver Perception of Change: X1 on Day 3
  • Clinician Global Impression of Change score: measures change in disease symptoms per clinician's judgement. Each item rated 1-7, 1=marked improvement, 7= marked worsening; min Caregiver perception of change interview: interviews with participants' caregiver(s). Open-ended questions elicit open-ended answers about subject's behavior, appearance, cognition, etc. over the study

OTHER OUTCOMES:
Pilot data on potential efficacy of PF 06412562 on individual domains of alertness | Once before and X2 after drug administration on Days 2 & 3
  Glasgow Coma scale (GCS): records consciousness; each item rated 1-6; score range: 3-14, where 3=deep unconsciousness, 15=totally alert Stanford Sleepiness Scale (SSS): measure of alertness; rated 1-7, 1=fully alert, 7=almost asleep, min total score=1, max total score=7
Pilot data on potential efficacy of PF 06412562 on individual domains of cogitation | Once before and X2 after drug administration on Days 2 & 3
  a. Severe Impairment Battery (SIB): evaluates cognition; min total score=0, max total score=100, higher score=lower cognition COGNISTAT: cognitive screening that assesses different domains of cognition Frontal Assessment Battery (FAB): used to assess different types of dementias. Min total score=0, max total score=18, higher scores=better performance
Pilot data on potential efficacy of PF 06412562 on individual domains of motor | Once before and X2 after drug administration on Days 2 & 3
  MDS-UPDRS-motor (III) (United Parkinson's Disease Rating Scale): each question scored on scale of 0 to 4, where 0= not present, 4= severe; min total score:0, max total score:81; higher score corresponds to increased disease severity
Pilot data on potential efficacy of PF 06412562 on individual domains of sleep | PSG sleep study: Days 1-3 at bedtime
  8 hour overnight polysomnography (PSG): sleep study monitoring body functions, brain activity (EEG), eye movements (EOG), muscle activity (EMG), and heart rhythm (ECG) Qualitative caregiver interview: (see outcome 2 description)

CONTACTS AND LOCATIONS:
Overall Officials: Xuemei Huang, MD, PhD, Principal Investigator — Milton S. Hershey Medical Center
Locations (1):
- Penn State Milton S. Hershey Medical Center, Hershey, Pennsylvania, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Fernandez-Mendoza J, Puzino K, Amatrudo G, Bourchtein E, Calhoun SL, Plante DT, Kaplan K. The Hypersomnia Severity Index: reliability, construct, and criterion validity in a clinical sample of patients with sleep disorders. J Clin Sleep Med. 2021 Nov 1;17(11):2249-2256. doi: 10.5664/jcsm.9426. PMID 34032202
- [Derived] Huang X, Lewis MM, Van Scoy LJ, De Jesus S, Eslinger PJ, Arnold AC, Miller AJ, Fernandez-Mendoza J, Snyder B, Harrington W, Kong L, Wang X, Sun D, Delnomdedieu M, Duvvuri S, Mahoney SE, Gray DL, Mailman RB. The D1/D5 Dopamine Partial Agonist PF-06412562 in Advanced-Stage Parkinson's Disease: A Feasibility Study. J Parkinsons Dis. 2020;10(4):1515-1527. doi: 10.3233/JPD-202188. PMID 32986682